CLINICAL TRIAL: NCT01072214
Title: A Randomized, Placebo-controlled, Double-masked, Parallel Group Study to Evaluate the Safety, Tolerability, and Pharmacokinetic Profile of Repeat Doses of Pazopanib Eye Drops in Healthy Adult Subjects
Brief Title: A Safety Study to Evaluate Pazopanib Eye Drops in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 113748
Record Dates: First submitted 2010-02-18; First posted 2010-02-22 (Estimated); Last update posted 2017-11-14 (Actual); Status verified 2017-11

CONDITIONS: Macular Degeneration
Keywords: Pazopanib; Tolerability; Pharmacokinetics; GW786034; Safety
MeSH Terms: conditions — Macular Degeneration | interventions — pazopanib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1.6 mg (Experimental): The actual dosage is 10 mg/ml (GW786034) given 4 times a day for a maximum daily dosage of 1.6mg
  Interventions: Drug: pazopanib
- TBD COHORT 2 (Experimental): Dose escalation amount to be determined (TBD) after results from Cohort 1 analyzed
  Interventions: Drug: pazopanib
- Placebo (Placebo Comparator): Subjects will receive placebo (drops without drug).
  Interventions: Drug: Placebo
- TBD COHORT 3 (Experimental): Dose escalation amount to be determined (TBD) after results from Cohort 2 analyzed
  Interventions: Drug: pazopanib

INTERVENTIONS:
Drug: pazopanib — gw786034
  Arms: TBD COHORT 2
Drug: pazopanib — gw786034
  Arms: 1.6 mg
Drug: pazopanib — gw786034
  Arms: TBD COHORT 3
Drug: Placebo — placebo
  Arms: Placebo

SUMMARY:
A study to determine the safety and tolerability of pazopanib eye drops. The study will also determine how the drug is absorbed and metabolized over time. Repeat doses of eye drops will be administered to healthy adult volunteers over a 14-day period with one additional dose given on the 15th day of the session. Three groups of subjects may receive either active drug or placebo (drops without drug). The first group of subjects will receive a maximum of 1.6mg of pazopanib or placebo. The dose of drug to be given to the next two groups will be determined based on the results of the first group of subjects. The last group of subjects will be of Japanese descent.

DETAILED DESCRIPTION:
The purpose of this study is to characterize the ocular safety and tolerability, the systemic safety and tolerability, and the pharmacokinetic profile of repeat doses of a higher strength ophthalmic formulation of pazopanib, 10 mg/mL. The higher strength formulation provides an opportunity to increase the total daily dose of pazopanib administered. In this 3-cohort study, healthy adult volunteers will participate in one 14-day repeat-dose session (plus a single dose on day 15), randomized to receive either pazopanib eye drops or placebo. Subjects in cohort 1 will receive 1 drop four times daily for a calculated total daily dose of 1.6 mg. The dosage regimen for two subsequent cohorts will be determined based on the emerging safety profile. The Japanese population chosen for the third cohort will provide a safety and tolerability profile as well as the pharmacokinetic profile of pazopanib prior to further development of this formulation in Japanese patients with AMD.

ELIGIBILITY:
Inclusion Criteria:

* AST, ALT, alkaline phosphatase and bilirubin ≤ 1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the Investigator and the GSK Medical Monitor agree that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Male or female ≥ 20 to 64 years of age, at the time of signing the informed consent.
* A female subject is eligible to participate if she is of non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea. In questionable cases, a blood sample with simultaneous follicle stimulating hormone (FSH) > 40 MlU/ml and estradiol < 40 pg/ml (<140 pmol/L) is confirmatory
* Body weight ≥ 50 kg for men and ≥ 45 kg for women and body mass index (BMI) within the range 18.5 - 32 kg/m2 (inclusive), where BMI = (weight in kg)/(height in meters)2.
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* Average QTcF < 450 msec or QTc < 480 msec in subjects with bundle branch block.
* Best-corrected visual acuity better than 20/80 (Snellen equivalent) in both eyes.

Exclusion Criteria:

* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* History of clinically relevant coronary heart disease, uncontrolled hypertension, renal disease, diabetes mellitus, impaired endocrine, thyroid, or respiratory function, or psychotic mental illness
* History of any hemorrhagic event (hemoptysis, cerebral or gastrointestinal) within 6 months of screening
* Urinary cotinine levels indicative of smoking or history or regular use of tobacco- or nicotine-containing products within 6 months of screening.
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening
* A positive pre-study drug/alcohol screen
* A positive test for HIV antibody
* Blood pressure (SBP/DBP) > 140/90 mmHg at screening
* History of dry eye or presence of any active ocular disease at time of screening that the investigator and medical monitor agree may cause additional risk to the subject or may interfere with study assessments or endpoints
* Any eye surgery within three months prior to first dose of study medication
* Use of ocular prescription or non-prescription drugs within 7 days prior to the first dose of study medication
* Prior history of ocular allergy, unless symptom-free for at least 6 months from first dose.
* An unwillingness to refrain from wearing contact lenses during the study and up to 2 weeks before the study start
* History of sensitivity to any of the study medications or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation
* History of regular alcohol consumption within 6 months of the study defined as:

an average weekly intake of >14 drinks for males or >7 drinks for females. One drink is equivalent to 12 g of alcohol: 12 ounces (360 mL) of beer, 5 ounces (150 mL) of wine or 1.5 ounces (45 mL) of 80-proof distilled spirits

* Participation in a clinical trial where the subject has received an investigational product within 30 days, 5 half-lives, or twice the duration of the biological effect of the investigational product (whichever is longer) prior to the first dose of study medication
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety
* Consumption of red wine, seville oranges, grapefruit or grapefruit juice within 7 days prior to the first dose of study medication
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period
* Unwillingness or inability to follow the procedures outlined in the protocol
* For Cohort 3, the following additional inclusion criterion applies:

Subject must have spent most of his or her life in Japan and not have lived outside of Japan for more than 5 years. They must have been born in Japan with four ethnic Japanese grandparents.

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2010-03-09 (Actual); Primary Completion 2010-06-28 (Actual); Study Completion 2010-06-28 (Actual)

PRIMARY OUTCOMES:
Clinical safety data from AE reporting, clinical observations, physical examinations, vital signs (blood pressure and heart rate), clinical laboratory tests including urinalysis, general ophthalmic examinations, and best-corrected visual acuity tests | 2 weeks
Primary pharmacokinetic endpoints will include: AUC(0-24), Cmax after repeat administration of pazopanib ophthalmic solution, Tmax, and trough steady-state plasma pazopanib concentration (Cτ) | 2 weeks

SECONDARY OUTCOMES:
Secondary pharmacokinetic parameters include: area under the plasma drug concentration versus time curve [AUC(0-t)], observed accumulation ratio (Ro), and apparent terminal half-life (t1/2) after repeat administration will be analyzed | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Glendale, California, United States

REFERENCES:
- [Derived] Singh R, Wurzelmann JI, Ye L, Henderson L, Hossain M, Trivedi T, Kelly DS. Clinical evaluation of pazopanib eye drops in healthy subjects and in subjects with neovascular age-related macular degeneration. Retina. 2014 Sep;34(9):1787-95. doi: 10.1097/IAE.0000000000000179. PMID 24896137
- See also: Results for study 113748 can be found on the GSK Clinical Study Register — https://www.gsk-clinicalstudyregister.com/study/113748?search=study&search_terms=113748#rs